CLINICAL TRIAL: NCT05432778
Title: Cytomegalovirus Prophylaxis With Letermovir in Heart Transplant Recipients: A Non-randomized Cohort Pilot Study
Brief Title: Cytomegalovirus Prophylaxis With Letermovir in Heart Transplant Recipients
Acronym: CYPHER-TXPilot
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 01
Record Dates: First submitted 2022-06-20; First posted 2022-06-27 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: CMV Viremia
Keywords: CMV reactivation; letermovir; heart transplantation
MeSH Terms: interventions — letermovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Group (Experimental): All patients in the Study Group will receive virostatic prophylaxis with letermovir 480 mg qd (We will be utilizing Letermovir oral formulation of 240 mg or 480 mg as available).
  Interventions: Drug: Letermovir Pill
- Control Group (No Intervention): Patients in Controls will receive standard-of-care virostatic prophylaxis with valgancyclovir 450 mg bid.

INTERVENTIONS:
Drug: Letermovir Pill — Patients in the Study Group will receive virostatic prophylaxis with letermovir 480 mg qd (We will be utilizing Letermovir oral formulation of 240 mg or 480 mg as available). n all patients the virostatic prophylaxis will be initiated between days 4 and 7 after heart transplantation and the duration of virostatic prophylaxis will be determined by the Quantiferon-CMV assay.
  Arms: Study Group

SUMMARY:
CMV infection is the most prevalent infection after heart transplantation (HTX), occurring in up to 40-60% of the recipients. It most frequently occurs within the first 6 months after transplantation and commonly presents as an asymptomatic viral replication. Viral syndrome or tissue-invasive disease (gastroenteritis, pneumonitis, myocarditis or meningitis) are much less common. Even though CMV infection is generally treatable with virostatic therapy and/or CMV-specific immunoglobulins, direct effects of CMV infection (viral syndrome and tissue-invasive disease) and general and transplant-specific indirect effects of CMV infection have been associated with significant morbidity and mortality in HTX patient population, mainly due to graft loss, development of malignancies, or opportunistic infections. According to the latest consensus paper on CMV prophylaxis and treatment in solid organ transplant recipients, valgancyclovir (or its active form gancyclovir) represents a virostatic therapy of choice for CMV prophylaxis and treatment after HTX. However, valgancyclovir has an array of side effects including hematological (leukopenia, neutropenia, anemia, thrombocytopenia), neurologic (headache, insomnia), gastrointestinal (decreased appetite, diarrhea, vomiting and dyspepsia) and psychiatric (depression) disorders. These can either expose HTX patients to additional complications (e.g. leukopenia and/or neutropenia can result in systemic fungal infections), decrease patients' quality of life, or mandate a decrease in valgancyclovir dose, which exposes patients to an increased risk for CMV reactivation. Recently, letermovir (a novel CMV viral terminase inhibitor), was approved for CMV prophylaxis in allogeneic bone marrow transplant recipients as the placebo-controlled study showed that significantly less patients, treated with letermovir, developed CMV disease (37% vs. 60%; P<0.001) and there was also a trend towards lower all-cause mortality. Data on bone marrow transplant recipients additionally suggest that letermovir is generally well tolerated with side effects limited to mild gastrointestinal symptoms (diarrhea, nausea). Importantly, myelosuppresive side effects of letermovir occur very rarely. Some encouraging data does exist on the use of letermovir in kidney transplant recipients, where a recently published proof-of-concept trial (N=27) suggested comparable safety and efficacy of leteremovir (N=18) and valgancyclovir (N=9): both treatment regimens resulted in similar time-course of viral load reduction and viral clearance and were well tolerated in terms of adverse events. Currently, a Phase III clinical trial is ongoing in renal transplant recipients (Clinicaltrials.gov: NCT03443869) to confirm this pilot data. However, to date, there is no published data on the use of letermovir in patients after HTX.

Based on the results in kidney transplantation, the aim of this pilot study is thus to evaluate the effects of letermovir-based CMV prophylaxis in heart transplant recipients.

The primary objective of the study is to investigate the efficacy of letermovir-based CMV prophylaxis in patients after heart transplantation.

The secondary objectives of the study are:

* to investigate the tolerability of letermovir-based CMV prophylaxis in patients after heart transplantation.
* to explore the potential correlation between letermovir-based CMV prophylaxis and restitution of cell-regulated immunity in patients after heart transplantation.

DETAILED DESCRIPTION:
This protocol represents a Phase II pilot prospective non-randomized single arm open-label study design. We aim to enroll 30 patients after heart transplantation (Study Group), who will meet all of the inclusion and none of the exclusion criteria and 60 propensity-matched historical controls (Controls; matched for gender, age, CMV serological status, CMV DNA quantification method, donor and transplant data and immunosuppresion treatment). All patients in the Study Group will receive virostatic prophylaxis with letermovir 480 mg qd (We will be utilizing Letermovir oral formulation of 240 mg or 480 mg as available). Patients in Controls will receive virostatic prophylaxis with valgancyclovir 450 mg bid. In all patients the virostatic prophylaxis will be initiated between days 4 and 7 after heart transplantation and the duration of virostatic prophylaxis will be determined by the Quantiferon-CMV assay. In all patients, initial Quantiferon-CMV assay evaluation will be performed 100 days post-heart transplant at which time PCR CMV assay will also be made. In patients with negative PCR CMV and Quantiferon-CMV values ≥ 0,2 IU/mL the virostatic therapy will be discontinued [10]. In patients with negative PCR CMV and Quantiferon-CMV values < 0,2 IU/mL the virostatic prophylaxis will continue for additional 30 days at which point Quantiferon-CMV assay will be re-evaluated. In an event of CMV infection/disease CMV it will be treated using valgancyclovir (900 mg q12) or gancyclovir (5 mg/kg q12h) per discretion of the treating heart transplant cardiologist and resistance to virostatic therapy will be tested at this time point. All patients (Study Group and Controls) will receive immunosuppresion induction therapy and triple maintenance immunosuppression therapy (TAC/MMF/steroid), fungal (posaconazole - 6 months), and pneumocystis prophylaxis (TMP/SMX - lifelong). In the Study Group additional, HSV /VZV viral prophylaxis with valacyclovir (500 mg q12, adjusted for renal function) will be used for 6 months after heart transplantation. Patients will be followed on an outpatient basis monthly for 12 months after enrollment and the events will be recorded using the following definitions. The maximum expected duration of letermovir therapy in the Study Group will be equal to the duration of follow-up - 12 months. After completion of the study all patients in the Study Group that may still require CMV virostatic prophylaxis according to our institutional guidelines will be switched to the current standard of care at our institution - valgancyclovir.

ELIGIBILITY:
Inclusion Criteria:

* heart transplant recipient (new)
* moderate (D+/R+ and D-/R+) or high (D+/R-) risk CMV serostatus
* signed informed consent for participation in the study

Exclusion Criteria:

* short-term mechanical circulatory support prior HTX
* ongoing CMV infection/disease
* D-/R- CMV serostatus
* heart re-transplantation
* need for intensified immunosuppression protocol

  * >20% cytolytic alloantibodies prior transplant
  * perioperative (within 7 days after HTX) allograft rejection > 1R
* immunoinduction with ATG
* pregnancy
* active participation in another interventional clinical trial
* know hypersensitivity to letermovir
* known hypersensitivity to valgancyclovir
* known hematological disorders (apart from anemia)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
The rate of early CMV infections/disease during virostatic prophylaxis. | baseline - 12 months
  The rate of early CMV infections/disease during virostatic prophylaxis.

SECONDARY OUTCOMES:
The rate of leukopenia during virostatic prophylaxis | baseline - 12 months
  The rate of leukopenia during virostatic prophylaxis
The rate of neutropenia during virostatic prophylaxis | baseline - 12 months
  The rate of neutropenia during virostatic prophylaxis
The rate of late CMV infections/disease between virostatic discontinuation and 6 months thereafter. | baseline - 12 months
  The rate of late CMV infections/disease between virostatic discontinuation and 6 months thereafter.
The time-course of the restitution of cell-mediated immunity during virostatic prophylaxis | baseline - 12 months
  The time-course of the restitution of cell-mediated immunity during virostatic prophylaxis
The rate of CMV resistance to virostatic therapy | baseline - 12 months
  The rate of CMV resistance to virostatic therapy

CONTACTS AND LOCATIONS:
Overall Officials: Bojan Vrtovec, MD, PhD, Principal Investigator — Advanced Heart Failure and Transplantation Center, Universtiy Medical Center Ljubljana, Slovenia
Locations (1):
- University Medical Center Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided